CLINICAL TRIAL: NCT06506526
Title: Clinical, Radiographical and Microbiological Evaluation of Chitosan as Irrigating Solution for Pulpectomy in Non-Vital Primary Teeth
Brief Title: Evaluation of Chitosan as Irrigating Solution for Pulpectomy in Non-Vital Primary Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: # 33/2017
Record Dates: First submitted 2024-03-16; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Pulpal Necrosis
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): The teeth will be irrigated by 2 ml 1% NaOCl after each file.
  Interventions: Procedure: Sodium hypochlorite irrigating solution
- One-minute NaOCL+Chitosan (Experimental): The teeth will be irrigated by 2 ml 1% NaOCl after each file then with 5 ml of 0.2% chitosan for one minute.
  Interventions: Procedure: one minute NaOCL+Chitosan
- Three-minute NaOCL+Chisosan (Experimental): The teeth will be irrigated by 2 ml 1% NaOCl after each file then with 5 ml of 0.2% chitosan for three minute.
  Interventions: Procedure: Three minute NaOCL+Chitosan

INTERVENTIONS:
Procedure: Sodium hypochlorite irrigating solution — 2 ml 1% NaOCl after each file
  Arms: Control group
Procedure: one minute NaOCL+Chitosan — 2 ml 1% NaOCl after each file then with 5 ml of 0.2% chitosan for one minute.
  Arms: One-minute NaOCL+Chitosan
Procedure: Three minute NaOCL+Chitosan — 2 ml 1% NaOCl after each file then with 5 ml of 0.2% chitosan for three minute.
  Arms: Three-minute NaOCL+Chisosan

SUMMARY:
45 teeth will be sub-divided at random with a computerized method, according to the type irrigant and duration of its application into 3 groups (15 teeth in each group):

Group1(control group):

The teeth will be irrigated by 2 ml 1% NaOCl after each file.

Group2:

The teeth will be irrigated by 2 ml 1% NaOCl after each file then with 5 ml of 0.2% chitosan for one minute.

Group 3:

The teeth will be irrigated by 2 ml 1% NaOCl after each file then with 5 ml of 0.2% chitosan for 3 minutes.

Evaluation

Clinical evaluation will be done for all groups at one, three, six and 12 months. The following parameters will be evaluated: Pain (spontaneous pain and pain with percussion) Degree of mobility Resolution of signs of infection (fistula) at the mucobuccal fold.

Radiographical evaluation will be performed to each patient immediately after the final restoration and three, six and 12 months postoperatively.

The decrease of radiolucency and the presence of internal or external root resorption will be evaluated.

Bacteriology :

The microbiological evaluation will be done at the Biotechnology Research Institute - Suez Canal University.

PCR will be used for detection of Enterococcus faecalis. Microbiological investigation will be used for counting the number of Enterococcus faecalis.

DETAILED DESCRIPTION:
45 teeth will be sub-divided at random with a computerized method, according to the type irrigant and duration of its application into 3 groups (15 teeth in each group):

Group1(control group):

The teeth will be irrigated by 2 ml 1% NaOCl after each file.

Group2:

The teeth will be irrigated by 2 ml 1% NaOCl after each file then with 5 ml of 0.2% chitosan for one minute.

Group 3:

The teeth will be irrigated by 2 ml 1% NaOCl after each file then with 5 ml of 0.2% chitosan for 3 minutes.

The root canals will then be flushed with 5 ml saline. Second microbiological sample will be collected. The tooth will be dried using paper points and then will be temporarily sealed with glass ionomer restoration.

Second Visit (after two days):

Glass ionomer will be removed and the third microbiological sample will be collected.

Zinc oxide and eugenol will be used as root canal filling material. All cases will be subjected to clinical and radiographical evaluation.

Evaluation

Clinical evaluation will be done for all groups at one, three, six and 12 months. The following parameters will be evaluated: Pain (spontaneous pain and pain with percussion) Degree of mobility Resolution of signs of infection (fistula) at the mucobuccal fold.

Radiographical evaluation will be performed to each patient immediately after the final restoration and three, six and 12 months postoperatively.

The decrease of radiolucency and the presence of internal or external root resorption will be evaluated.

Bacteriology :

The microbiological evaluation will be done at the Biotechnology Research Institute - Suez Canal University.

PCR will be used for detection of Enterococcus faecalis. Microbiological investigation will be used for counting the number of Enterococcus faecalis.

Microbiological sample collection protocol:

Two sterile paper points will be introduced into the canals until they reached the full working length, and kept in place for 60 seconds (19). Each paper point will be immediately embedded in 3ml sterile tube containing adequate transporting medium or saline solution.

The first tube will be transported to the microbiological laboratory for culturing within a maximum of 2 hours, while the other tube will be kept at -80 °C for DNA extraction and direct detection of Enterococcus faecalis via multiplex PCR assay.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy Children aged from three to seven years.
* No previous history of antibiotics for at least two weeks.
* Non- Vital primary teeth that can be fully isolated.
* Presence of clinical signs or symptoms suggesting a non-vital tooth, such as intra-oral fistula.
* Infection diagnosed by presence of periapical radiolucency in a periapical radiograph.
* Root resorption not more than one third of the root.
* Patient and parent cooperation.

Exclusion Criteria:

* Non-restorable tooth
* Serious reduction in bone support and/or extreme tooth mobility.
* Radiographic indication of extensive internal or external root resorption.

Ages: 3 Months to 7 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Spontanous Pain | after one month, 3 months, six months and 12 months
  Visual analog scale "A scale from 1 to 10 where 1 is mild pain and 10 Worst pain"
Radiographical evaluation | immediately after restoration, 3 months, six months and 12 months
  The change of radiolucency
Radiographic examination " internal or external root resorption" | immediately after restoration, 3 months, six months and 12 months
  Presence (1) or absence (0)
Bacteriology | During procedure
  PCR will be used for detection of Enterococcus faecalis.
  - Microbiological investigation will be used for counting the number of Enterococcus faecalis

CONTACTS AND LOCATIONS:
Locations (1):
- Mostafa youssef, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No